CLINICAL TRIAL: NCT05719246
Title: Standardized Yoga & Meditation Program for Stress Reduction for Adolescents With Irritable Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-126
Record Dates: First submitted 2022-03-07; First posted 2023-02-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Irritable Bowel Syndrome; Anxiety; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS Patients Doing Yoga (Experimental): All patients will fall under the arm of "IBS Patients Doing Yoga" and will follow the yoga videos that are assigned to them during the study. The participants are their own controls and their symptom changes will be recorded pre- and post-video watching and participation.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — The yoga video set that the participants will follow is a brief, at-home, 6-week twice per week Standardized Yoga & Meditation Program for Stress Reduction (SYMPro-SR) program. The videos feature Sydney Topfer guiding the participants through different yoga poses.

SUMMARY:
Irritable Bowel Syndrome (IBS) is the most common cause of recurrent abdominal pain in children. IBS is a functional gastrointestinal disorder that is linked to motor and sensory physiology, as well as the central nervous system, that presents as abdominal pain with abnormal defecation patterns. This discomfort leads to emotional stress, decreased quality of life, and anxiety. The study proposes that yoga and mindfulness will decrease anxiety and increase quality of life for patients with IBS. The aim of this study is to measure the impact of a brief, at-home, 6-week twice per week Standardized Yoga & Meditation Program for Stress Reduction program on anxiety, IBS symptoms, and quality of life in children ages 12-21 diagnosed with IBS.

DETAILED DESCRIPTION:
Background: Irritable Bowel Syndrome (IBS), is the most common cause of general recurrent abdominal pain (RAP) in children. IBS is a functional gastrointestinal disorder that is linked to motor and sensory physiology, as well as the central nervous system, that presents as abdominal pain with abnormal defecation patterns. This discomfort often significantly impacts the patient's life, leading to emotional stress, decreased quality of life due to necessary changes in daily living to accommodate bathroom patterns, as well as anxiety and depression. Since IBS is often accompanied by anxiety, along with other psychological and quality of life issues, it will be evaluated whether practicing yoga and mindfulness will decrease anxiety and increase quality of life for patients with IBS

Objective: To measure the impact of a brief, at-home, 6-week twice per week Standardized Yoga & Meditation Program for Stress Reduction (SYMPro-SR) program on anxiety, IBS symptoms, and quality of life in children ages 12-21 years old diagnosed with Irritable Bowel Syndrome.

Methods: This is a pilot, IRB approved, prospective study. Children ages 12-21 who suffer from any of the four types of Irritable Bowel Syndromes will be identified. Each subject will be asked to fill out the Screen for Child Anxiety Related Disorders, Children Somatic Symptoms Inventory and Pediatric Quality of Life Inventory questionnaires before and after an online, 6- week yoga course. Anxiety will be measured using the Screen for Child Anxiety Related Disorders and quality of life will be measured using Pediatric Quality of Life Inventory and Children Somatic Symptoms Inventory tests. Results of the questionnaires total scores and sub-scales will be analyzed as continuous variables using paired t-tests or the Wilcoxon signed rank tests for the pre-post results and ANCOVA for repeated measures incorporating age, sex, baseline scores, etc. as covariates. Comparisons within the group will be done using Student paired t-test for continuous data. The difference will be considered significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Cooper Pediatric Gastroenterology practice in Camden, NJ or Voorhees, NJ
* Patients of Cooper Pediatric Gastroenterology practice in Voorhees, NJ
* Participants 12 to 21 years old with any type of IBS diagnosis
* Subjects must be able to access the internet to be able to watch the yoga videos on Youtube
* Patients must complete 4 out of 6 modules to stay in the study

Exclusion Criteria:

* Participants under the age of 12
* Participants over the age of 21

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life | Change from Pre intervention to 6 weeks after intervention (at completion of intervention which lasts 6 weeks)
  Pediatric Quality of Life Inventory questionnaire will be used
Children Somatic Symptoms Inventory | Change from Pre intervention to 6 weeks after intervention (at completion of intervention which lasts 6 weeks)
  Children Somatic Symptoms Inventory questionnaire will be used
Anxiety | Change from Pre intervention to 6 weeks after intervention (at completion of intervention which lasts 6 weeks)
  Screen for Child Anxiety Related Disorders questionnaire will be used

CONTACTS AND LOCATIONS:
Overall Officials: Alla Kushnir, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chumpitazi BP, Self MM, Czyzewski DI, Cejka S, Swank PR, Shulman RJ. Bristol Stool Form Scale reliability and agreement decreases when determining Rome III stool form designations. Neurogastroenterol Motil. 2016 Mar;28(3):443-8. doi: 10.1111/nmo.12738. Epub 2015 Dec 21. PMID 26690980
- [Background] Lacy BE, Patel NK. Rome Criteria and a Diagnostic Approach to Irritable Bowel Syndrome. J Clin Med. 2017 Oct 26;6(11):99. doi: 10.3390/jcm6110099. PMID 29072609
- [Background] Locke GR 3rd, Pemberton JH, Phillips SF. AGA technical review on constipation. American Gastroenterological Association. Gastroenterology. 2000 Dec;119(6):1766-78. doi: 10.1053/gast.2000.20392. PMID 11113099
- [Background] Khalsa SB, Hickey-Schultz L, Cohen D, Steiner N, Cope S. Evaluation of the mental health benefits of yoga in a secondary school: a preliminary randomized controlled trial. J Behav Health Serv Res. 2012 Jan;39(1):80-90. doi: 10.1007/s11414-011-9249-8. PMID 21647811
- [Background] Huguet A, Izaguirre Eguren J, Miguel-Ruiz D, Vall Valles X, Alda JA. Deficient Emotional Self-Regulation in Children with Attention Deficit Hyperactivity Disorder: Mindfulness as a Useful Treatment Modality. J Dev Behav Pediatr. 2019 Jul/Aug;40(6):425-431. doi: 10.1097/DBP.0000000000000682. PMID 31135603
- [Background] Evans S, Seidman LC, Lung K, Sternlieb B, Zeltzer LK. Yoga for Teens With Irritable Bowel Syndrome: Results From a Mixed-Methods Pilot Study. Holist Nurs Pract. 2018 Sep/Oct;32(5):253-260. doi: 10.1097/HNP.0000000000000288. PMID 30113959
- [Background] Devanarayana NM, Rajindrajith S. Irritable bowel syndrome in children: Current knowledge, challenges and opportunities. World J Gastroenterol. 2018 Jun 7;24(21):2211-2235. doi: 10.3748/wjg.v24.i21.2211. PMID 29881232
- [Background] Reigada LC, Hoogendoorn CJ, Walsh LC, Lai J, Szigethy E, Cohen BH, Bao R, Isola K, Benkov KJ. Anxiety symptoms and disease severity in children and adolescents with Crohn disease. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):30-5. doi: 10.1097/MPG.0000000000000552. PMID 25187105
- [Result] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05719246/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT05719246/ICF_001.pdf